CLINICAL TRIAL: NCT02848612
Title: Evaluation of the Amiens University Hospital Neuroradiology Anticoagulation Protocol
Acronym: ANTICONEURORAD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2015-13 Pr Lorne
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Aneurysm
Keywords: anticoagulation; aneurysmal subarachnoid haemorrhage; interventional neuroradiology; coil embolization
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: anticoagulation by unfractionated heparin — anticoagulation by unfractionated heparin

SUMMARY:
To prevent thromboembolic complications, the embolization procedure is performed under prophylactic unfractionated heparin, the efficacy of which is monitored by point-of- care testing according to international guidelines. However, these guidelines are based on limited scientific evidence and the ideal level of anticoagulation required has not been precisely defined. Furthermore, the correlation between the point-of- care tests used at Amiens University Hospital and the reference methods used in the laboratory varies considerably according to the available literature.

DETAILED DESCRIPTION:
Since the beginning of the 2000s, the reference treatment for the management of aneurysmal subarachnoid haemorrhage consists of interventional neuroradiology with coil embolization of the aneurysm. Although ensuring a better neurological prognosis than neurosurgical clipping, interventional neuroradiology exposes the patient to various risks: thromboembolic complications during or after embolization and re-rupture of the aneurysm during embolization. To prevent thromboembolic complications, the embolization procedure is performed under prophylactic unfractionated heparin, the efficacy of which is monitored by point-of- care testing according to international guidelines. However, these guidelines are based on limited scientific evidence and the ideal level of anticoagulation required has not been precisely defined. Furthermore, the correlation between the point-of- care tests used at Amiens University Hospital and the reference methods used in the laboratory varies considerably according to the available literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years undergoing one of the following interventional neuroradiology procedures at Amiens University Hospital: elective embolization of an intracranial aneurysm, emergency embolization of a ruptured intracranial aneurysm, elective or urgent embolization of an intracranial or perispinal arteriovenous malformation.

Exclusion Criteria:

* Patients in whom all modalities of monitoring of the efficacy of anticoagulation (laboratory tests and point-of-care tests) were not performed, incomplete embolization or radiological follow-up records.
* Patients presenting a contraindication to the administration of unfractionated heparin: history of heparin-induced thrombocytopenia or haemorrhagic coagulopathy (von Willebrand disease, haemophilia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 years undergoing one of the following interventional neuroradiology procedures at Amiens University Hospital: elective embolization of an intracranial aneurysm, emergency embolization of a ruptured intracranial aneurysm, elective or urgent embolization of an intracranial or perispinal arteriovenous malformation.
Sampling Method: Non-Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
correlation between laboratory clotting tests and point-of-care clotting tests | 6 months
  evaluation of the correlation between laboratory clotting tests and point-of-care clotting tests performed on the Hemochron Junior® device.
  care clotting tests and laboratory tests in the setting of intracranial
  embolization.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel LORNE, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France